CLINICAL TRIAL: NCT02955537
Title: MI-BP: mHealth to Improve Blood Pressure Control
Acronym: MI-BP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: Wayne State University (Other); Vanderbilt University (Other); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Lorraine Buis, Associate Professor of Family Medicine, Medical School and Associate Professor of Information, School of Information, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HUM00114202; 1R01HL127215-01A1 (NIH)
Record Dates: First submitted 2016-11-02; First posted 2016-11-04 (Estimated); Last update posted 2023-03-01 (Actual); Status verified 2023-02

CONDITIONS: Hypertension
Keywords: Hypertension; mHealth
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual care (No Intervention): Usual care participants will be given a prescription for antihypertensive medications, printed educational materials on hypertension, and a home blood pressure monitor for daily use, but will receive no further intervention.
- MI-BP (Experimental): MI-BP participants will receive an antihypertensive medication prescription, and be asked to use technology-mediated devices/services linked to positive changes in target behavior/outcome including the MI-BP app, a secure, mHealth platform that will be installed on participant smartphones.
  Interventions: Other: MI-BP

INTERVENTIONS:
Other: MI-BP — MI-BP includes the following components: 1) Home blood pressure monitoring 2) Physical activity monitoring 3) Sodium intake self-monitoring 4) Physical activity and sodium intake goal setting 5) Educational messaging via push notification and in-app messaging 6) motivational messaging 7) tailored messaging relevant to individual participants and 8) medication reminders.
  Arms: MI-BP

SUMMARY:
This study seeks to evaluate a multicomponent mobile intervention to change multiple hypertension-related health behaviors in minorities and the underserved with uncontrolled hypertension. Half of the participants will receive a mobile intervention designed to improve physical activity, sodium intake, and medication adherence. The other half will receive usual care.

ELIGIBILITY:
Inclusion Criteria:

* Detroit-area residents
* Hypertensive
* Owning a compatible smartphone
* Presenting to the Detroit Medical Center Detroit Receiving, Sinai-Grace Hospital, or selected Community Health Screening Events with, but not necessarily for, uncontrolled blood pressure (systolic blood pressure ≥ 135 mm Hg at triage and on repeat measurement using the BpTRU device).

Exclusion Criteria:

* No self-reported prior history of hypertension
* No hypertension diagnosis documented in their medical record
* Non-English speaking
* Presenting with an acute illness necessitating immediate medical intervention
* Presenting with an admission to the hospital for critical reasons (as determined by the attending physician)
* Pregnant (as determined by a dip test at screening), or self-report during trial.
* Having the following serious comorbidities or confounders due to the fact that they may make blood pressure control difficult or necessitate frequent Emergency Department use or hospitalization:

  * Previous diagnosis of resistant hypertension (or current use of 3 or more maximally dosed antihypertensive agents without achievement of blood pressure control)
  * Steroid dependent asthma or emphysema
  * Cirrhosis or hepatic failure
  * Chronic heart failure (any stage)
  * Previous diagnosis of acute myocardial infarction, angina (stable or unstable), or known coronary artery disease
  * Previous diagnosis of cerebrovascular disease (including transient ischemic attack or stroke)
  * Known valvular heart disease
  * Stage IV or V chronic kidney disease
  * Cancer (terminal or undergoing active chemotherapeutic or radiation therapy)
* Patients with other serious medical conditions that may affect their ability to self-monitor blood pressure (such a dementia)
* Having a history of alcohol or drug abuse as determined by the CAGE-AID questionnaire (excluded if 2 or more)
* Week 2 measurement of systolic blood pressure < 130 mm Hg using the BpTRU device or study-issued BP cuff.

Ages: 25 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 162 (Actual)
Dates: Start 2018-01-11 (Actual); Primary Completion 2021-04-15 (Actual); Study Completion 2021-04-15 (Actual)

PRIMARY OUTCOMES:
Change in mean systolic blood pressure | from baseline to 1 year

SECONDARY OUTCOMES:
Change in physical activity as measured by the International Physical Activity Questionnaire (IPAQ-SF) | from baseline to 1 year
Change in sodium intake as measured by the Block Sodium Screener | from baseline to 1 year
Change in medication adherence as measured by Adherence to Refills and Medications Scale (ARMS) | from baseline to 1 year
Change in blood pressure control | from baseline to 1 year

OTHER OUTCOMES:
Cost-effectiveness of MI-BP compared to usual care | within-trial
Cost-effectiveness of MI-BP compared to usual care | long-term

CONTACTS AND LOCATIONS:
Overall Officials: Lorraine R Buis, PhD, Principal Investigator — University of Michigan
Locations (2):
- United States (2):
  - University of Michigan, Ann Arbor, Michigan
  - Wayne State University, Detroit, Michigan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Buis LR, Kim J, Sen A, Chen D, Dawood K, Kadri R, Muladore R, Plegue M, Richardson CR, Djuric Z, McNaughton C, Hutton D, Robert LP, Park SY, Levy P. The Effect of an mHealth Self-Monitoring Intervention (MI-BP) on Blood Pressure Among Black Individuals With Uncontrolled Hypertension: Randomized Controlled Trial. JMIR Mhealth Uhealth. 2024 Jun 28;12:e57863. doi: 10.2196/57863. PMID 38941601